CLINICAL TRIAL: NCT05333263
Title: Validation of Treadmill Disturbance Parameters
Brief Title: A Study to Validate Treadmill Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenton R. Kaufman, PhD, PE, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-007581; W81XWH-20-C-0104 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- ABB Motor (Experimental): Subjects will undergo a balance assessment using the following program on the treadmill: 3-phase-motor, velocity control mode.
  Interventions: Device: Treadmetrix
- ETM Motor (Experimental): Subjects will undergo a balance assessment using the following program on the treadmill: single-phase, velocity control mode.
  Interventions: Device: Treadmetrix
- NIDEC/CT Motor (Experimental): Subjects will undergo a balance assessment using the following program on the treadmill: single-phase motor, position-mode.
  Interventions: Device: Treadmetrix

INTERVENTIONS:
Device: Treadmetrix — Programmable treadmill that delivers controlled postural disturbances

SUMMARY:
The purpose of this study is to evaluate the accuracy with which a microprocessor-controlled treadmill delivers controlled postural disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with no medical conditions or previous injuries, trauma, or surgeries that reduce your balance, mobility or strength.
* Able to follow simple directions.
* Willingness to participate in the study.
* No restriction will be placed on gender, race, or ethnicity.

Exclusion Criteria:

* Current or chronic pain in your shoulders, elbows, hips, knees, ankles, feet, neck or back.
* Use of assistive device such as walker or cane.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenton Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ABB Motor: Subjects underwent a balance assessment using the following program on the treadmill: 3-phase motor, velocity-control mode.
  Treadmetrix: Programmable treadmill that delivers controlled postural disturbances
- ETM Motor: Subjects will undergo a balance assessment using the following program on the treadmill: single-phase, velocity control mode.
  Device: Treadmetrix Programmable treadmill that delivers controlled postural disturbances
- NIDEC/CT Motor: Subjects will undergo a balance assessment using the following program on the treadmill: single-phase motor, position-mode.
  Device: Treadmetrix Programmable treadmill that delivers controlled postural disturbances
Period: Overall Study
Arm/Group | ABB Motor | ETM Motor | NIDEC/CT Motor
Started | 5 | 2 | 5
Completed | 5 | 2 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABB Motor | ETM Motor | NIDEC/CT Motor | Total
Number analyzed (Participants) | 5 | 2 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 5 | 12
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 4 | 1 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Limits of Agreement Between Observed and Commanded Treadmill Belt Disturbance Parameters: Belt Displacement.
Description: Treadmill belt displacement (cm) will be measured with a Motion Capture system for each perturbation trial and compared to the commanded magnitude to assess system accuracy. Mean observed treadmill belt displacement, in centimeters, relative to commended treadmill belt displacement was calculated and the mean relative error (percentage) was reported. Percent Error = (Commanded Kinematic Value - Observed Kinematic Value)/Commanded Kinematic Value *100%. The mean value is then determined from the individual errors for each participant. This results in Mean Relative Error. Lower numbers are considered a better outcome (less error). A negative percentage indicates that the observed value is larger than the command value.
Time Frame: Duration of participant test session (approximately 2 hours)
Measure: Mean (Standard Deviation); unit: Mean Relative Error (%)
Arm/Group | ABB Motor | ETM Motor | NIDEC/CT Motor
Number analyzed (Participants) | 5 | 2 | 5
Mean Relative Error (%)
  4 cm | -8.5 (4.2) | 20.0 (1.3) | 2.1 (1.2)
  20 cm | -5.8 (0.5) | -6.6 (0.8) | -0.2 (0.1)
  40 cm | -5.9 (0.4) | -7.5 (2.3) | -0.5 (0.1)
  60 cm | -6.0 (0.9) | -2.9 (0.7) | -3.1 (2.8)
  80 cm | -3.8 (1.4) | 9.4 (0.6) | -2.4 (3.9)
  -4 cm | -2.8 (2.9) | 20.0 (3.0) | 2.2 (1.2)
  -20 cm | -5.5 (0.3) | -6.9 (2.2) | -0.3 (0.3)
  -40 cm | -5.6 (0.4) | -2.6 (6.0) | -0.6 (0.2)
  -60 cm | -5.0 (0.4) | 5.1 (2.8) | -0.8 (0.5)
  -80 cm | -2.0 (2.8) | 16.8 (3.0) | 3.1 (1.1)

2. Primary Outcome: Estimate the Limits of Agreement Between Observed and Commanded Treadmill Belt Disturbance Parameters: Peak Velocity.
Description: Treadmill belt peak velocity (cm/s) will be measured with a Motion Capture system for each perturbation trial and compared to the commanded magnitude to assess system accuracy. Mean observed treadmill belt peak velocity, in centimeters/second, relative to commended treadmill belt peak velocity was calculated and the mean relative error (percentage) was reported. Percent Error = (Commanded Kinematic Value - Observed Kinematic Value)/Commanded Kinematic Value *100%. The mean value is then determined from the individual errors for each participant. This results in Mean Relative Error. Lower numbers are considered a better outcome (less error). A negative percentage indicates that the observed value is larger than the command value.
Time Frame: Duration of participant test session (approximately 2 hours)
Measure: Mean (Standard Deviation); unit: Mean Relative Error (%)
Arm/Group | ABB Motor | ETM Motor | NIDEC/CT Motor
Number analyzed (Participants) | 5 | 2 | 5
Mean Relative Error (%)
  20 cm/s | 0.1 (0.5) | 15.8 (3.2) | -0.9 (0.8)
  100 cm/s | -2.9 (0.8) | -2.9 (4.0) | -2.1 (0.9)
  200 cm/s | -3.9 (0.5) | -5.8 (2.0) | -2.7 (0.9)
  300 cm/s | -3.3 (0.4) | 4.3 (2.6) | -1.0 (0.7)
  400 cm/s | -2.5 (0.4) | 20.4 (1.1) | 14.4 (2.0)
  -20 cm/s | 1.7 (1.6) | 15.4 (1.8) | -0.2 (1.4)
  -100 cm/s | -1.7 (1.2) | 0.8 (1.0) | -1.8 (1.2)
  -200 cm/s | -2.5 (0.6) | 2.2 (2.5) | -2.3 (1.5)
  -300 cm/s | -2.7 (0.6) | 11.6 (0.2) | 0.1 (1.0)
  -400 cm/s | -0.8 (1.1) | 27.2 (0.8) | 17.3 (2.3)

3. Primary Outcome: Estimate the Limits of Agreement Between Observed and Commanded Treadmill Belt Disturbance Parameters: Average Initial Acceleration.
Description: Treadmill belt average initial acceleration (cm/s/s) will be measured with a Motion Capture system for each perturbation trial and compared to the commanded magnitude to assess system accuracy. Mean observed treadmill belt average initial acceleration, in centimeters/second/second, relative to commended treadmill belt average initial acceleration was calculated and the mean relative error (percentage) was reported. Percent Error = (Commanded Kinematic Value - Observed Kinematic Value)/Commanded Kinematic Value *100%. The mean value is then determined from the individual errors for each participant. This results in Mean Relative Error. Lower numbers are considered a better outcome (less error). A negative percentage indicates that the observed value is larger than the command value.
Time Frame: Duration of participant test session (approximately 2 hours)
Measure: Mean (Standard Deviation); unit: Mean Relative Error (%)
Arm/Group | ABB Motor | ETM Motor | NIDEC/CT Motor
Number analyzed (Participants) | 5 | 2 | 5
Mean Relative Error (%)
  100 cm/s/s | 0.2 (7.4) | -6.9 (0.7) | -15.2 (4.7)
  500 cm/s/s | 1.1 (3.5) | 5.8 (1.6) | -1.6 (1.1)
  1000 cm/s/s | 1.7 (1.5) | 5.9 (3.0) | -0.5 (0.9)
  1500 cm/s/s | 1.8 (0.8) | 18.7 (3.0) | 2.4 (1.2)
  2000 cm/s/s | 3.0 (1.2) | 37.3 (2.6) | 25.3 (3.1)
  -100 cm/s/s | -2.8 (6.5) | -7.2 (1.3) | -14.9 (6.4)
  -500 cm/s/s | 2.6 (1.4) | 8.7 (3.6) | -0.4 (1.9)
  -1000 cm/s/s | 3.4 (0.8) | 15.9 (5.2) | 0.6 (2.3)
  -1500 cm/s/s | 2.4 (0.5) | 29.8 (1.0) | 4.6 (1.9)
  -2000 cm/s/s | 5.9 (2.2) | 45.8 (0.1) | 28.0 (3.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 2 hours.
Arm/Group | ABB Motor | ETM Motor | NIDEC/CT Motor
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT05333263/Prot_001.pdf